CLINICAL TRIAL: NCT04273581
Title: The Efficacy and Safety of Thalidomide Combined With Low-dose Hormones in the Treatment of Severe New Coronavirus (COVID-19) Pneumonia: a Prospective, Multicenter, Randomized, Double-blind, Placebo, Parallel Controlled Clinical Study
Brief Title: The Efficacy and Safety of Thalidomide Combined With Low-dose Hormones in the Treatment of Severe COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other); Wenzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200214-COVID-19-S-T
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: COVID-19 Thalidomide
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): α-interferon： nebulized inhalation, 5 million U or equivalent dose added 2ml of sterile water for injection, 2 times a day, for 7 days； Abidol, 200mg / time, 3 times a day, for 7 days; Methylprednisolone： 40mg, q12h， for 5 days. placebo：100mg/d，qn，for 14 days.
  Interventions: Drug: placebo
- Thalidomide group (Experimental): α-interferon： nebulized inhalation, 5 million U or equivalent dose added 2ml of sterile water for injection, 2 times a day, for 7 days； Abidol, 200mg / time, 3 times a day, for 7 days; Methylprednisolone： 40mg, q12h， for 5 days. thalidomide：100mg/d，qn，for 14 days.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: placebo — 100mg/d，qn，for 14 days.
  Arms: Control group
Drug: Thalidomide — 100mg/d，qn，for 14 days.
  Other Names: fanyingting
  Arms: Thalidomide group

SUMMARY:
In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of lung injury caused by COVID-19 can be an alternative target for current treatment. Patients with severe COVID-19 have rapid disease progression and high mortality. There is currently no effective treatment method, which may be related to the excessive immune response caused by cytokine storm. This study will evaluate thalidomide combined with low-dose hormone adjuvant therapy for severe COVID-19 Patient effectiveness and safety.

DETAILED DESCRIPTION:
Thalidomide has been clinically reported, and combined with antiviral drugs and other conventional treatments have achieved good results in the treatment of severe H1N1, especially after the death of a young severe patient. After the addition of thalidomide, the reported 35 patients did not Deaths. Subsequent basic research at Fudan University confirmed that thalidomide can treat H1N1 lung injury. And think that the combination with antiviral drugs may be a better alternative strategy for H1N1 before the vaccine is successfully developed.

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of lung injury caused by COVID-19 can be an alternative target for current treatment. Patients with severe COVID-19 have rapid disease progression and high mortality. There is currently no effective treatment method, which may be related to the excessive immune response caused by cytokine storm.It has been reported that the combined use of thalidomide and dexamethasone can effectively inhibit NK / T-cell lymphoma combined with ECSIT V140A mutation of hematophilic syndrome. The AIDS immune reconstitution syndrome (IRIS) is also an abnormal inflammatory response in nature. It has been reported that thalidomide as an immunomodulatory agent for the treatment of IRIS is effective. This study will evaluate thalidomide combined with low-dose hormone adjuvant therapy for severe COVID-19 Patient effectiveness and safety.

Although the death rate of COVID-19 infected persons is not high, their rapid infectiousness and the lack of effective antiviral treatment currently have become the focus of the national and international epidemic. Thalidomide has been available for more than sixty years, and has been widely used in clinical applications. It has been proved to be safe and effective in IPF, severe H1N1 influenza lung injury and paraquat poisoning lung injury, and the mechanism of anti-inflammatory and anti-fibrosis is relatively clear. As the current research on COVID-19 at home and abroad mainly focuses on the exploration of antiviral efficacy, this study intends to find another way to start with host treatment in the case that antiviral is difficult to overcome in the short term, in order to control or relieve lung inflammation caused by the virus To improve lung function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. The laboratory (RT-PCR) confirmed the diagnosis of severe patients infected with CoVID-19 (refer to the fifth edition of the Chinese diagnosis and treatment guideline for trial); the diagnosis of new coronavirus pneumonia was confirmed, and any of the following: 1) Respiratory distress, breathing ≥30 beats / min; 2) In the resting state, the oxygen saturation is ≤93%; 3) Arterial blood oxygen partial pressure / oxygen concentration ≤300mmHg
3. The diagnosis is less than or equal to 12 days;

Exclusion Criteria:

1. Severe liver disease (such as Child Pugh score ≥ C, AST> 5 times the upper limit); severe renal dysfunction (the glomerulus is 30ml / min / 1.73m2 or less)
2. Pregnancy or breastfeeding or positive pregnancy test;
3. In the 30 days before the screening assessment, have taken any experimental treatment drugs for CoVID-19 (including off-label, informed consent use or trial-related);
4. Those with a history of thromboembolism, except for those caused by PICC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-18 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Improvement (TTCI) | up to 28 days
  TTCI is defined as the time (in days) from initiation of study treatment (active or placebo) until a decline of two categories from admission status on a six-category ordinal scale of clinical status which ranges from 1 (discharged) to 6 (death). Six-category ordinal scale: 6. Death; 5. ICU, requiring ECMO and/or IMV; 4. ICU/hospitalization, requiring NIV/ HFNC therapy; 3. Hospitalization, requiring supplemental oxygen (but not NIV/ HFNC); 2. Hospitalization, not requiring supplemental oxygen; 1. Hospital discharge. Abbreviation: IMV, invasive mechanical ventilation; NIV, non-invasive mechanical ventilation; HFNC, High-flow nasal cannula.

SECONDARY OUTCOMES:
Clinical status | days 7, 14, 21, and 28
  Clinical status, assessed by the ordinal scale at fixed time points
Time to Hospital Discharge OR NEWS2 (National Early Warning Score 2) of ≤ 2 maintained for 24 hours | up to 28 days
All cause mortality | up to 28 days
Duration (days) of mechanical ventilation | up to 28 days
Duration (days) of extracorporeal membrane oxygenation | up to 28 days
Duration (days) of supplemental oxygenation | up to 28 days
Length of hospital stay (days) | up to 28 days
Time to 2019-nCoV RT-PCR negativity in upper and lower respiratory tract specimens | up to 28 days
Change (reduction) in 2019-nCoV viral load in upper and lower respiratory tract specimens as assessed by area under viral load curve. | up to 28 days
Frequency of serious adverse drug events | up to 28 days
Serum TNF-α, IL-1β, IL-2, IL-6, IL-7, IL-10, GSCF, IP10#MCP1, MIP1α and other cytokine expression levels before and after treatment | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinglin Xia, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University

REFERENCES:
- [Background] Jin YH, Cai L, Cheng ZS, Cheng H, Deng T, Fan YP, Fang C, Huang D, Huang LQ, Huang Q, Han Y, Hu B, Hu F, Li BH, Li YR, Liang K, Lin LK, Luo LS, Ma J, Ma LL, Peng ZY, Pan YB, Pan ZY, Ren XQ, Sun HM, Wang Y, Wang YY, Weng H, Wei CJ, Wu DF, Xia J, Xiong Y, Xu HB, Yao XM, Yuan YF, Ye TS, Zhang XC, Zhang YW, Zhang YG, Zhang HM, Zhao Y, Zhao MJ, Zi H, Zeng XT, Wang YY, Wang XH; , for the Zhongnan Hospital of Wuhan University Novel Coronavirus Management and Research Team, Evidence-Based Medicine Chapter of China International Exchange and Promotive Association for Medical and Health Care (CPAM). A rapid advice guideline for the diagnosis and treatment of 2019 novel coronavirus (2019-nCoV) infected pneumonia (standard version). Mil Med Res. 2020 Feb 6;7(1):4. doi: 10.1186/s40779-020-0233-6. PMID 32029004
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Background] Bartlett JB, Dredge K, Dalgleish AG. The evolution of thalidomide and its IMiD derivatives as anticancer agents. Nat Rev Cancer. 2004 Apr;4(4):314-22. doi: 10.1038/nrc1323. No abstract available. PMID 15057291
- [Background] Zhao L, Xiao K, Wang H, Wang Z, Sun L, Zhang F, Zhang X, Tang F, He W. Thalidomide has a therapeutic effect on interstitial lung fibrosis: evidence from in vitro and in vivo studies. Clin Exp Immunol. 2009 Aug;157(2):310-5. doi: 10.1111/j.1365-2249.2009.03962.x. PMID 19604271
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wen H, Ma H, Cai Q, Lin S, Lei X, He B, Wu S, Wang Z, Gao Y, Liu W, Liu W, Tao Q, Long Z, Yan M, Li D, Kelley KW, Yang Y, Huang H, Liu Q. Recurrent ECSIT mutation encoding V140A triggers hyperinflammation and promotes hemophagocytic syndrome in extranodal NK/T cell lymphoma. Nat Med. 2018 Feb;24(2):154-164. doi: 10.1038/nm.4456. Epub 2018 Jan 1. PMID 29291352
- [Background] Zhu H, Shi X, Ju D, Huang H, Wei W, Dong X. Anti-inflammatory effect of thalidomide on H1N1 influenza virus-induced pulmonary injury in mice. Inflammation. 2014 Dec;37(6):2091-8. doi: 10.1007/s10753-014-9943-9. PMID 24912813
- [Background] Kwon HY, Han YJ, Im JH, Baek JH, Lee JS. Two cases of immune reconstitution inflammatory syndrome in HIV patients treated with thalidomide. Int J STD AIDS. 2019 Oct;30(11):1131-1135. doi: 10.1177/0956462419847297. Epub 2019 Sep 19. No abstract available. PMID 31533530
- See also: Clinical characteristics of 2019 novel coronavirus infection in China by Nan-Shan Zhong — http://doi.org/10.1101/2020.02.06.20020974